CLINICAL TRIAL: NCT00121329
Title: 4% Intrauterine Lidocaine Infusion for Pain Management in First Trimester Abortions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB 6876
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2005-07-21 (Estimated); Status verified 2005-07

CONDITIONS: Pain
Keywords: Pain with procedures
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Intrauterine lidocaine infusion 4%

SUMMARY:
Recent studies have investigated the use of local anesthetics (i.e. lidocaine, mepivacaine) to lessen the pain experienced with minor gynecologic procedures such as endometrial biopsy and office hysteroscopy. Local anesthetic injected into the uterine cavity has been demonstrated effective in some studies at decreasing patient pain associated with these intrauterine procedures at an anesthetic concentration of at least 2%. Based on this evidence, we hypothesized that an intrauterine lidocaine infusion may reduce patient pain during first trimester abortions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Good general health
* English speaking
* Confirmation of gestational age by ultrasound
* Body weight > 100 lbs.
* Pregnancy < 11 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2004-12

PRIMARY OUTCOMES:
VAS scores during cervical dilation and uterine aspiration

SECONDARY OUTCOMES:
Patient satisfaction, symptoms, lidocaine levels

CONTACTS AND LOCATIONS:
Overall Officials: Alison B Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Planned Parenthood of the Columbia Willamette, Portland, Oregon, United States